CLINICAL TRIAL: NCT01758562
Title: Caphosol® Versus State-of-the-art Mouthcare in Patients With Allogeneic Stem Cell Transplantation: a Randomized Controlled Study About the Efficacy of the Mouth Rinse Caphosol®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Capo
Record Dates: First submitted 2012-12-24; First posted 2013-01-01 (Estimated); Last update posted 2014-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Allogeneic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- State-of-the-art mouth care (No Intervention)
- Mouth rinse Caphosol (Active Comparator): Mouth rinse,aqueous solution. Caphosol is a preparation comprising two separately packaged aqueous solutions, a phosphate solution and a calcium solution, which, when both solutions are combined in equal volumes, forms a solution supersaturated with respect to both calcium and phosphate ions.
  Interventions: Device: Caphosol

INTERVENTIONS:
Device: Caphosol
  Arms: Mouth rinse Caphosol

SUMMARY:
Randomized controlled study about the efficacy of the mouth rinse Caphosol in patients with allogeneic stem cell transplantation. 85% of the patients receive a severe oral mucositis due to their treatment.

70 patients will be randomized in the intervention (Caphosol) or in the standard (state-of-the-art) group. Primary endpoint is the duration of the mucositis, secondary endpoints are the occurence of oral mucositis measured with the WHO-scale and the occurence of pain measured with the NRS-scale (Numeric Rating Scale).

* Trial with medical device

ELIGIBILITY:
Inclusion criteria:

* Allogeneic stem cell transplantation
* Male and female patients age 18-80
* Signed informed consent after information

Exclusion criteria:

* Contra-indications due to ethical reasons
* Unable to read or write
* Unable to speak or understand the german language
* Low-salt diet

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2013-01; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Duration of oral mucositis | 20-30 days

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Spirig, Prof MD, Principal Investigator — University Hospital Zurich, Centre of Clinical Nursing Science
Locations (1):
- University Hospital Zurich, Centre of Clinical Nursing Science, Zurich, Canton of Zurich, Switzerland